CLINICAL TRIAL: NCT01558544
Title: Cryopreservation of Ovarian Tissue for Potential In Vitro Maturation or Autologous Transplantation
Brief Title: Cryopreservation of Ovarian Tissue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0901010165
Record Dates: First submitted 2012-02-16; First posted 2012-03-20 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-10

CONDITIONS: Cancer; Risk of Premature Ovarian Failure; Fertility Preservation
Keywords: Ovarian tissue cryopreservation; Ovarian tissue transplantation; Fertility preservation; Risk of premature ovarian failure
MeSH Terms: conditions — Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use of high dose chemotherapy (Other): Use of chemotherapy without removal of the disease ovary.
  Interventions: Procedure: surgery to remove ovaries or high dose chemotherapy

INTERVENTIONS:
Procedure: surgery to remove ovaries or high dose chemotherapy — oophorectomy to remove a disease ovary.
  Other Names: Use of high dose chemotherapy without removal of disease ovary.

SUMMARY:
The study hopes to contribute to the development of technologies of ovarian tissue freezing-thawing and in vitro maturation of immature eggs such that a person at risk for premature ovarian failure might be able to conceive a genetically related child.

DETAILED DESCRIPTION:
Procedure: The patient will undergo preoperative sonographic assessment of both ovaries to determine if either ovary is diseased or compromised. Patient will undergo preoperative blood sampling to measure AMH, FSH, LH and estradiol as indicators of current ovarian function (less than 8 teaspoons) if time allows and assessment of ovarian reserve is appropriate; menopausal levels of FSH (≥ 30 miu/ml) will be a contraindication to participation in this study. The patient may have infectious disease testing as part of the evaluation for fertility preservation treatment. Patient will undergo preoperative assessment and clearance for surgery by an anesthesiologist.

Intraoperative management will include laparotomy or laparoscopy, depending on the individual patient's history, exam and oncology plans. Removal of one or both ovaries will depend on preoperative ovarian assessment and recommendation of the oncologist. If ovarian survival for the anticipated treatment has never been documented then both ovaries will be removed. Both ovaries may also be removed if diseased or if the condition requires prophylactic oophorectomy to prevent risk of malignant transformation, e.g. 46 XX/46 XY chimera and BRCA mutation carriers. If ovarian function has rarely been documented for the anticipated treatment then one ovary will be removed and one may be left in situ or repositioned to avoid the field of radiation. The decision to leave the ovary in situ or to reposition will be made pre-operatively by the physician performing the surgery in consultation with the patient and the radiation oncologist. If there is no normal ovarian tissue, as determined by pathology, we will take biopsies of ovarian tissue not to exceed 50% of the ovarian volume from the contra-lateral side for freezing. Additionally, the remaining ovary may be repositioned and sutured to the posterior wall of the uterus or above the pelvic brim with a radio-opaque clip placed to identify this ovary for shielding during irradiation.

Ovarian tissue will be removed and treated as follows: (a) the cortex will be stripped from the remaining ovarian tissue as this outer layer contains most of the immature eggs or primordial follicles. The cortex will be sectioned into 8mm x 1mm strips, each to be frozen in vials containing 1-3 strips. One strip will be sent to pathology for paraffin embedding to be available for future assessment of occult lymphoma cells markers; (b) the central or medullary portion will be frozen separately for potential scientific analysis since this section would not be of any clinical utility. The amount of tissue frozen may vary depending in part by whether one or two ovaries are removed. At some point in the future, thawing of ovarian tissue, with either in vitro maturation or autologous transplantation into the pelvis or other area of the body could be performed. The patient would receive routine postoperative care. The patient's oncologist will be consulted regarding proper timing of the surgery and the need for any special intraoperative or postoperative management

However, since the survival of the primordial follicles in transplanted ovarian tissue is quite low (<10%), methods for in vivo maturation of these eggs and improved methods of transplantation need to be developed. One or two vials of tissue (<10% of all tissue frozen) will be thawed to develop the techniques of maturing oocytes. This may include transplantation of the tissue into an animal model for in vivo maturation.

Six months to 1 year following surgery and/or treatment for the medical condition, eg chemotherapy, hormone testing will be performed for evaluation of ovarian reserve. This may include AMH and FSH hormone levels as well as pelvic ultrasounds and dominant antra follicle count.

If the subject does not wish to utilize the ovarian tissue for her own clinical use, the options include discarding the cryopreserved ovarian tissue or donating the cryopreserved tissue for approved research studies.

ELIGIBILITY:
Inclusion Criteria:

* Females 0-45 years of age who are premenopausal
* Treatment plan that will likely result in premature menopause or premature ovarian failure
* This includes patients receiving:
* Cancer treatment with abdominal pelvic irradiation and/or high dose chemotherapy
* Surgery that requires removal of ovaries for medical condition or disease, e.g. Prophylactic oophorectomy in BRCA patients
* Patient is unable or unwilling to pursue fertility preservation by freezing oocytes or embryos.
* Previous treatment for cancer is acceptable if patient still has ovarian function
* Patient is medically stable enough to undergo surgery (cleared for anesthesia)

Exclusion Criteria:

* Patients not meeting the above criteria
* Patients who have not received medical clearance from their physicians to undergo surgery
* Patients already experiencing menopause.

Max Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Estimated)
Dates: Start 1997-04 (Actual); Primary Completion 2029-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
CRYOPRESERVATION OF OVARIAN TISSUE FOR POTENTIAL IN VITRO MATURATION OR AUTOLOGOUS TRANSPLANTATION | 6 months to a year post surgery, hormone testing will be performed to test ovarian function.
  Ovarian tissue cryopreservation Survival of tissue undergoing cryopreservation, thawing and maturation of immature eggs.

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Schattman, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Ronald O. Perelman and Claudia Cohen Center for Reproductive Medicine, New York, New York, United States